CLINICAL TRIAL: NCT01906749
Title: Colchicine for Acute Coronary Syndromes. A Multicenter Double Blind Randomized Trial.
Brief Title: Colchicine for Acute Coronary Syndromes
Acronym: COACS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Vittoria Hospital (Other)
Responsible Party: Principal Investigator, Massimo Imazio, MD, Maria Vittoria Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27/06/13; 2013-001415-78 (EudraCT Number)
Record Dates: First submitted 2013-07-21; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Colchicine
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Colchicine (Active Comparator): Colchicine 0.5mg once daily for 24 months
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — 0.5mg once daily orally
  Arms: Colchicine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Multicenter, double blind, randomized trial to assess the effect of low-dose colchicine (0.5mg/day) on overall mortality, new coronary syndromes, and ischemic stroke at 2 years after an acute coronary syndrome. The study hypothesis is that colchicine may reduce the specified combined endpoint from 16% to 7-8% at a 2-years follow-up.

DETAILED DESCRIPTION:
Multicenter, double-blind randomized trial to evaluate the efficacy of low dose colchicine (0.5mg once daily for 2 years) to reduce the incidence of subsequent overall mortality, new acute coronary syndromes, and ischemic stroke in patients admitted for an acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* >18years
* Acute coronary syndrome (unstable angina or acute myocardial infarction)
* Life expectancy> 2 years
* Absence of contraindications to colchicine

Exclusion Criteria:

* Colchicine treatment for any cause
* Severe liver disease
* Renal insufficiency with creatinine>150mmol/l or creatinine clearance<30ml/min/1.73m2
* Known cancer
* Chronic inflammatory bowel disease
* treatment with cyclosporine
* allergy or hypersensitivity to colchicine
* pregnancy or lactating woman or woman with childbearing potential without valid contraception

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Overall mortality, new acute coronary syndrome, and ischemic stroke. | 24 months

SECONDARY OUTCOMES:
Mortality | 24 months
  Secondary outcome measures will contain each issue of the combined primary endpoint as separate outcome.
New acute coronary syndrome (unstable angina and myocardial infarction) | 24 months
Ischemic Stroke | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Imazio, MD, Study Chair — Cardiology Dpt.Maria Vittoria Hospital, Torino, Italy
Locations (3):
- Italy (3):
  - Cardiology Dpt., Rivoli, Torino
  - Cardiology Dpt.Maria Vittoria Hospital, Torino, Torino
  - Cardiology Dpt.San Giovanni Bosco Hospital, Torino, Torino

REFERENCES:
- [Derived] Silvis MJM, Demkes EJ, Fiolet ATL, Dekker M, Bosch L, van Hout GPJ, Timmers L, de Kleijn DPV. Immunomodulation of the NLRP3 Inflammasome in Atherosclerosis, Coronary Artery Disease, and Acute Myocardial Infarction. J Cardiovasc Transl Res. 2021 Feb;14(1):23-34. doi: 10.1007/s12265-020-10049-w. Epub 2020 Jul 9. PMID 32648087